CLINICAL TRIAL: NCT06798480
Title: Prevalence of Problematic Use of Social Media in the General PopuLation
Brief Title: Prevalence of Problematic Use of Social Media
Acronym: PURPLE
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0042; 2024-A02539-38 (Other: ID-RCB)
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Social Networks; Addiction
Keywords: Problematic use; social media; addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Social media users: All French individuals aged 13 years or older who use social media
  Interventions: Other: Self-administered survey

INTERVENTIONS:
Other: Self-administered survey — An anonymous self-administered online questionnaire hosted on LimeSurvey, lasting approximately 20 minutes, will be completed by participants. A panel of participants representative of the general population will be provided by the Selvitys Institute. In parallel, the self-administered questionnaire will also be distributed via posts on social media platforms (Facebook, YouTube, Instagram, TikTok, Snapchat, and X) over a period of three months.

SUMMARY:
In 2023, French individuals spend an average of two hours per day on social media platforms (SM), primarily Facebook, TikTok, X, YouTube, Instagram, and Snapchat. While social media offers undeniable benefits, it also raises concerns about its impact on mental health and well-being. These impacts remain poorly understood, partly due to the diversity of social media uses and motivations, which do not have uniform effects on health. For instance, studies have shown that "active" use of social media (e.g., content creation) is associated with higher well-being, whereas "passive" use (e.g., content scrolling) is linked to lower well-being.

This challenge in understanding the variety of social media uses and their consequences has direct clinical implications. Clinicians working in pediatrics, child psychiatry, and addiction medicine are increasingly confronted with patients struggling to manage their social media use. However, they lack clear diagnostic criteria to differentiate between normal and problematic use, as well as specific tools tailored to address potential disorders.

Moreover, in France, there is no existing estimate of the proportion of the general population affected by problematic social media use.

This study aims to establish the prevalence of problematic use of social media in France. The investigators hypothesize that the prevalence will be close to 10%, which is the prevalence that has been found in other European countries in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 years or older.
* Resident in France and French-speaking.
* Does not object to participating in the study, and, for minors, whose parents also do not object to their participation.

Exclusion Criteria:

* Unable to understand and complete the questionnaire (e.g., non-French-speaking).

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Panel population (probability sample):The first study population will consist of a panel of 3,900 participants provided by the Selvitys Institute. These participants are selected using probability sampling methods to ensure that they are representative of the general French population aged 13 years or older. The selection is based on key demographic characteristics such as age, gender, and geographic location, level of education, ensuring a diverse and balanced sample.
  Social media population (non-probability sample):The second study population will consist of individuals who voluntarily respond to the online self-administered questionnaire through recruitment campaigns on social media platforms. This non-probability sample is composed of individuals who actively use social media and are interested in participating. As participation is voluntary, the sample may not fully represent the broader French population but will provide insights into social media users' behavior and experiences
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of problematic use of social media. | baseline
  Outcome measure: Problematic use will be identified if the participant endorses at least 6 out of 9 items on the French version of the Social Media Addiction Scale. The prevalence of problematic use will be calculated as the number of participants with problematic use divided by the total number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Julia DE TERNAY, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France